CLINICAL TRIAL: NCT06462807
Title: Improving the Organizational Social Context to Address Structural Racism and Discrimination: A Randomized Controlled Trial to Reduce Racial Disparities in Viral Suppression and Retention in HIV Care
Brief Title: Improving the Organizational Social Context to Address Structural Racism and Discrimination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Florence Momplaisir, MD, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-38
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accessibility, Responsiveness, Continuity (ARC) (Experimental)
  Interventions: Behavioral: ARC
- Standard of Care (SOC) (No Intervention)

INTERVENTIONS:
Behavioral: ARC — ARC is an evidence-based intervention that uses three strategies (ARC principles, ARC component tools, and ARC mental models) to create organizational social contexts (OSCs) that support the implementation of interventions to improve patient outcomes.
  Arms: Accessibility, Responsiveness, Continuity (ARC)

SUMMARY:
Despite the widespread use of effective antiretroviral therapy (ART), the HIV epidemic continues to impact racial and ethnic minority populations disproportionately. Although Black/African American persons account for 13% of the U.S. population, they account for 41% of new HIV diagnoses and experience the lowest rates of retention in HIV care and viral suppression (VS) compared to other racial/ethnic groups. Structural racism and discrimination (SRD) likely contribute to racial disparities in HIV outcomes.

Although the outpatient setting is a vitally important aspect of care provision for people living with HIV (PLWH), there are limited data on the impact of intra-organizational SRD on HIV outcomes. Longitudinal engagement in HIV care is needed for sustained VS and decreased community transmission of HIV. The organizational social context (OSC) includes organizational culture (organizational norms and values that drive quality of care), organizational climate (perception of the culture and how it impacts personal well-being), and workers' attitudes. Using a randomized controlled trial (RCT), we will implement ARC (Accessibility, Responsiveness, Continuity) to improve organizational behavior and reduce racial disparities in HIV outcomes for PLWH. ARC is an evidence-based intervention that uses three strategies (ARC principles, ARC component tools, and ARC mental models) to create OSCs that support the implementation of interventions to improve patient outcomes.

Clinics will be randomized to ARC (n = 2) or standard of care (SOC; n= 2). Those assigned to ARC will address SRD occurring at the organizational level affecting care, including referral and treatment patterns for PLWH. A pre-implementation period will be followed by ARC and ARC-associated implementation strategies for 36 months and then a 12-month post-implementation period where we will continue to measure HIV outcomes in both arms. We will compare HIV outcomes, namely VS and retention in care, and intermediate outcomes, such as linkage to mental health treatment and staff turn-over in clinics assigned to ARC and SOC.

We will also evaluate whether individual (self-efficacy, perceived discrimination) and organizational factors (OSC and cohesion of OSC measures) mediate the relationship between ARC, intermediate, and HIV outcomes. In preparation to the RCT, we will evaluate baseline OSC measures across 12 HIV clinics in Philadelphia and determine aspects of the OSC associated with VS and retention in care in a multi-level model adjusting for neighborhood SRD, patient-level factors, and clustering of patients nested in clinics and neighborhoods. We will then test the effectiveness of ARC in improving a primary outcome of VS and secondary outcome of retention in care at the end of the implementation period. We will examine the acceptability, sustainability, and cost of implementing ARC in outpatient HIV care. This research will advance understanding of the impact of SRD on HIV treatment outcomes and health services research and the implementation of a disseminable evidence-based practice aimed at reducing SRD.

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

* PLWH: in care in one of 12 clinics in Philadelphia

  1. HIV diagnosis date at least one year prior to the administration of the clinic OSC measures
  2. Philadelphia address at the time of HIV diagnosis
  3. successfully linked to care at any point during the study period, defined as having documentation of 1 or more CD4 or Viral Load test results after the date of diagnosis
* Clinic workers: clinic leaders, administrators, frontline staff, and providers across participating clinics

Aim 2:

* PLWH: having an established diagnosis of HIV and receiving care at one of the 4 clinics at least 6 months before the pre-implementation period
* Clinic workers: the entire pool of workers employed in the 2 clinics assigned to the intervention arm will be invited to participate in ARC

Aim 3:

- Clinic staff and PLWH at clinics receiving ARC

Exclusion Criteria:

Aim 1:

* PLWH: Persons in a correctional facility will be excluded from this analysis
* Clinic workers: Participants who are not employed in one of the roles that were designated

Aim 2:

* PLWH: Patients who get discharged from a clinic because they moved (or for other reasons) or who died will not be eligible to enter the pre-implementation cohort.
* Clinic workers: Clinics assigned to SOC will not receive ARC but will be asked to complete surveys using the same schedule as the clinics assigned to receive ARC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Viral Suppression | 12-month period
  HIV-1 RNA <400 copies per milliliter

SECONDARY OUTCOMES:
Retention in HIV Care | 12-month period
  defined as at least 1 medical visit with a provider with prescribing privileges in each 6-month interval of the 12-month measurement period, with a minimum of 60 days between medical visits

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States